CLINICAL TRIAL: NCT05574491
Title: Comparative Effectiveness of Traditional and Computerized Versions of the Transdiagnostic Program Super Skills for Life in Children Aged 8-12 Years: a Randomized Controlled Trial
Brief Title: Effectiveness of Traditional and Computerized Versions of Super Skills for Life in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 220118115011
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Depressive Disorder; Depressive Symptoms; Anxiety Disorders; Anxiety Disorders and Symptoms; Mood Disorders; Emotional Disorder
MeSH Terms: conditions — Depressive Disorder; Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants who met the inclusion criteria and underwent thorough the baseline assessment will be randomly assigned to the conditions of the intervention groups (traditional and computerized versions of SSL).
  Children allocated to the traditional and multimedia versions of the SSL program will receive the eight-week intervention.
  Participants in WLC group will receive no psychological intervention during the eight-week duration of the program.
  Children and parents in the three groups will complete the same series of measures at about the same time (pre-test and after eight weeks). Children in WLC group will receive the intervention once the follow-up visit is completed.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Super Skills for Life intervention group: traditional version (Experimental): The Super Skills for Life program will be administered following the manual of the intervention by a trained therapist, as described in the section of intervention/treatment.
  Interventions: Behavioral: Super Skills for Life: traditional version
- Super Skills for Life intervention group: computerized version (Experimental): The Super Skills for Life program will be administered in-person as well by a trained therapist, as described in the section of intervention treatment.
  The therapist will use the multimedia presentation of the program's contents as a tool for the better development of the sessions. The digital version of the program consists of an animation whose characters narrate examples that help the children better understand the contents. The therapist will have a password assigned to each child, and it will be the therapist who will guide the sessions and select the contents of the digital presentation that correspond to each session. The web address to access the programme is https://www.superskillsonline.com/.
  Interventions: Behavioral: Super Skills for Life: computerized version

INTERVENTIONS:
Behavioral: Super Skills for Life: traditional version — Structured and manualized intervention with a manual for the therapist and a workbook for the children.
  The intervention will be administered by trained clinical psychologists in SSL. Sessions will be held once a week for eight weeks, with each session lasting approximately forty five minutes.
  The program includes emotional education, social skills training, cognitive restructuring, relaxation techniques, self-observation, problem solving and behavioural activation. These contents are learned through playful exercises, activities, readings, and role-playing.
  Both modalities of intervention will be in-person.
  Spanish version of Super Skills for Life group program: Orgilés, M., Espada, J.P., Ollendick, T.H. & Essau, C. (2022). Programa Super Skills. Manual del aplicador. Elche, ES: Universidad Miguel Hernández.
  Arms: Super Skills for Life intervention group: traditional version
Behavioral: Super Skills for Life: computerized version — Structured and manualized intervention with a manual for the therapist and multimedia material for the children.
  Arms: Super Skills for Life intervention group: computerized version

SUMMARY:
Super Skills for Life (SSL) is a transdiagnostic cognitive-behavioral protocol developed for children aged 6 to 12 with anxiety and comorbid problems (e.g., depression, low self-esteem, and lack of social skills).

SSL consists of eight sessions targeting common risk factors for internalizing disorders such as cognitive distortions, avoidance, emotional management, low self-esteem, social skills deficits and coping strategies.

The aim of the study is to investigate the comparative effectiveness of SSL in its traditional and computerized versions on internalizing symptoms in Spanish children between 8 and 12 years of age.

DETAILED DESCRIPTION:
Children will be selected to receive the SSL program based on results on psychometrically robust measurements and inclusion/exclusion criteria. Selected children will be randomly assigned to the conditions of the two intervention groups (traditional and computerized versions of SSL).

Parents and children from the two groups will complete the same measures at baseline and post-treatment. They will also complete these measures at 6 months follow-up, and 12 months follow-up.

Researchers will compare the results of pre-test to post-test assessments in children participating in the traditional and multimedia versions of SSL on depressive symptoms, anxiety symptoms, interference of anxiety on child's life, self-esteem, social skills, social worries, and cognitive emotional regulation.

The investigators will also assess these variables in the intervention group at 6 months and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 - 12 years old.
* Presence of emotional symptoms, which will be assessed using the SCAS and the MFQ, parent versions. The cut-off point for inclusion in the study is a score equal to or above 25 on the SCAS and/or equal to or above 20 on the MFQ.
* Speaking, reading, writing and understanding Spanish.

Exclusion Criteria:

* Intellectual disability, behavioral symptoms, or autism spectrum symptoms whose severity precluded continued treatment.
* Being receiving current psychological or pharmacological treatment for anxiety and/or depression.
* Not accepting or revoking informed consent to participate in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline children's reported anxiety symptoms | Baseline
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms immediately after the intervention | Immediately after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms at 6 months | 6 months after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms at 12 months | 12 months after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Baseline parent-reported anxiety symptoms | Baseline
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms immediately after the intervention | Immediately after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms immediately at 6 months | 6 months after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms immediately at 12 months | 12 months after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Baseline children's reported depressive symptoms | Baseline
  Measured by Mood and Feelings Questionnaire - Short Version (MFQS). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Children's reported depressive symptoms immediately after the intervention | Immediately after the intervention
  Measured by Mood and Feelings Questionnaire - Short Version (MFQS). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Children's reported depressive symptoms at 6 months | 6 months after the intervention
  Measured by Mood and Feelings Questionnaire - Short Version (MFQS). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Children's reported depressive symptoms at 12 months | 12 months after the intervention
  Measured by Mood and Feelings Questionnaire - Short Version (MFQS). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Baseline parent-reported depressive symptoms | Baseline
  Measured by Mood and Feelings Questionnaire Parent-Report (MFQ-P). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 68). Higher scores indicate more severe symptoms.
Parent-reported depressive symptoms immediately after the intervention | Immediately after the intervention
  Measured by Mood and Feelings Questionnaire Parent-Report (MFQ-P). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 68). Higher scores indicate more severe symptoms.
Parent-reported depressive symptoms immediately at 6 months | 6 months after the intervention
  Measured by Mood and Feelings Questionnaire Parent-Report (MFQ-P). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 68). Higher scores indicate more severe symptoms.
Parent-reported depressive symptoms immediately at 12 months | 12 months after the intervention
  Measured by Mood and Feelings Questionnaire Parent-Report (MFQ-P). It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 68). Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Baseline children's anxiety-related interference | Baseline
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Children's anxiety-related interference immediately after the intervention | Immediately after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Children's anxiety-related interference at 6 months | 6 months after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Children's anxiety-related interference at 12 months | 12 months after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Baseline parent-reported anxiety-related interference | Baseline
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference immediately after the intervention | Immediately after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference at 6 months | 6 months after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference at 12 months | 12 months after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Baseline self-esteem | Baseline
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem immediately after the intervention | Immediately after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem at 6 months | 6 months after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem at 12 months | 12 months after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Baseline social skills | Baseline
  Social Skills Questionnaire (SSQ). It measures children's social functioning, as reflected by specific behavioural responses during interaction with another person. The scale consists of 30 items rated 0 to 2 points. Minimum value 0 and maximum value 60. Higher scores indicate higher social skills.
Social skills immediately after the intervention | Immediately after the intervention
  Social Skills Questionnaire (SSQ). It measures children's social functioning, as reflected by specific behavioural responses during interaction with another person. The scale consists of 30 items rated 0 to 2 points. Minimum value 0 and maximum value 60. Higher scores indicate higher social skills.
Social skills at 6 months | 6 months after the intervention
  Social Skills Questionnaire (SSQ). It measures children's social functioning, as reflected by specific behavioural responses during interaction with another person. The scale consists of 30 items rated 0 to 2 points. Minimum value 0 and maximum value 60. Higher scores indicate higher social skills.
Social skills at 12 months | 12 months after the intervention
  Social Skills Questionnaire (SSQ). It measures children's social functioning, as reflected by specific behavioural responses during interaction with another person. The scale consists of 30 items rated 0 to 2 points. Minimum value 0 and maximum value 60. Higher scores indicate higher social skills.
Baseline social worries | Baseline
  Social Worries Questionnaire (SSW). It measures children's social worries, in terms of anxiety about and avoidance of specific social situations in which social evaluation or scrutiny by others is likely to occur. The scale consists of 12 items rated 0 to 2 points. Minimum value 0 and maximum value 24. Higher scores indicate higher social worries.
Social worries immediately after the intervention | Immediately after the intervention
  Social Worries Questionnaire (SSW). It measures children's social worries, in terms of anxiety about and avoidance of specific social situations in which social evaluation or scrutiny by others is likely to occur. The scale consists of 12 items rated 0 to 2 points. Minimum value 0 and maximum value 24. Higher scores indicate higher social worries.
Social worries at 6 months | 6 months after the intervention
  Social Worries Questionnaire (SSW). It measures children's social worries, in terms of anxiety about and avoidance of specific social situations in which social evaluation or scrutiny by others is likely to occur. The scale consists of 12 items rated 0 to 2 points. Minimum value 0 and maximum value 24. Higher scores indicate higher social worries.
Social worries at 12 months | 12 months after the intervention
  Social Worries Questionnaire (SSW). It measures children's social worries, in terms of anxiety about and avoidance of specific social situations in which social evaluation or scrutiny by others is likely to occur. The scale consists of 12 items rated 0 to 2 points. Minimum value 0 and maximum value 24. Higher scores indicate higher social worries.
Baseline cognitive emotion regulation strategies | Baseline
  Measured by the Cognitive Emotion Regulation Questionnaire (CERQ-k). CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Cognitive emotion regulation strategies immediately after the intervention | Immediately after the intervention
  Measured by the Cognitive Emotion Regulation Questionnaire children self-report (CERQ-k). CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Cognitive emotion regulation strategies at 6 months | 6 months after the intervention
  Measured by the Cognitive Emotion Regulation Questionnaire children self-report (CERQ-k). CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Cognitive emotion regulation strategies at 12 months | 12 months after the intervention
  Measured by the Cognitive Emotion Regulation Questionnaire children self-report (CERQ-k). CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Baseline parental depression, anxiety and stress symptoms | Baseline
  Measured by the Depression Anxiety Stress Scales - short version (DASS-21). It contains a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Baseline parental depression, anxiety and stress symptoms | Immediately after the intervention
  Measured by the Depression Anxiety Stress Scales - short version (DASS-21). It contains a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Baseline parental depression, anxiety and stress symptoms | 6 months after the intervention
  Measured by the Depression Anxiety Stress Scales - short version (DASS-21). It contains a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.
Baseline parental depression, anxiety and stress symptoms | 12 months after the intervention
  Measured by the Depression Anxiety Stress Scales - short version (DASS-21). It contains a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Orgilés Amorós, Principal Investigator — Miguel Hernandez University of Elche
Locations (1):
- Department of Health Psychology. Miguel Hernandez University of Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting after finishing all analysis and publication.
Access Criteria: Upon request and verification by the principal investigator to consult the available data. The use of the data for distribution in any format is not permitted.

REFERENCES:
- [Background] Essau CA, Olaya B, Sasagawa S, Pithia J, Bray D, Ollendick TH. Integrating video-feedback and cognitive preparation, social skills training and behavioural activation in a cognitive behavioural therapy in the treatment of childhood anxiety. J Affect Disord. 2014;167:261-7. doi: 10.1016/j.jad.2014.05.056. Epub 2014 Jun 4. PMID 24999861
- [Background] Essau CA, Sasagawa S, Jones G, Fernandes B, Ollendick TH. Evaluating the real-world effectiveness of a cognitive behavior therapy-based transdiagnostic program for emotional problems in children in a regular school setting. J Affect Disord. 2019 Jun 15;253:357-365. doi: 10.1016/j.jad.2019.04.036. Epub 2019 Apr 16. PMID 31078836
- [Background] Orgiles M, Fernandez-Martinez I, Espada JP, Morales A. Spanish version of Super Skills for Life: short- and long-term impact of a transdiagnostic prevention protocol targeting childhood anxiety and depression. Anxiety Stress Coping. 2019 Nov;32(6):694-710. doi: 10.1080/10615806.2019.1645836. Epub 2019 Jul 23. PMID 31334667
- [Background] Fernandez-Martinez I, Orgiles M, Morales A, Espada JP, Essau CA. One-Year follow-up effects of a cognitive behavior therapy-based transdiagnostic program for emotional problems in young children: A school-based cluster-randomized controlled trial. J Affect Disord. 2020 Feb 1;262:258-266. doi: 10.1016/j.jad.2019.11.002. Epub 2019 Nov 4. PMID 31733917
- [Background] Melero S, Orgiles M, Espada JP, Morales A. Spanish version of Super Skills for Life in individual modality: Improvement of children's emotional well-being from a transdiagnostic approach. J Clin Psychol. 2021 Oct;77(10):2187-2202. doi: 10.1002/jclp.23148. Epub 2021 Apr 21. PMID 33882156
- [Background] Fernandez-Martinez I, Morales A, Espada JP, Orgiles M. Effects of Super Skills for Life on the social skills of anxious children through video analysis. Psicothema. 2020 May;32(2):229-236. doi: 10.7334/psicothema2019.240. PMID 32249749
- [Background] Melero S, Morales A, Espada JP, Mendez X, Orgiles M. Effectiveness of Group vs. Individual Therapy to Decrease Peer Problems and Increase Prosociality in Children. Int J Environ Res Public Health. 2021 Apr 9;18(8):3950. doi: 10.3390/ijerph18083950. PMID 33918640
- [Background] Melero S, Morales A, Espada JP, Orgiles M. Improving Social Performance Through Video-feedback with Cognitive Preparation in Children with Emotional Problems. Behav Modif. 2022 Jul;46(4):755-781. doi: 10.1177/0145445521991098. Epub 2021 Jan 29. PMID 33511861
- [Background] Escribano S, Espada JP, Orgiles M, Morales A. Implementation fidelity for promoting the effectiveness of an adolescent sexual health program. Eval Program Plann. 2016 Dec;59:81-87. doi: 10.1016/j.evalprogplan.2016.08.008. Epub 2016 Aug 31. PMID 27614301
- [Background] Orgiles M, Melero S, Fernandez-Martinez I, Espada JP, Morales A. Effectiveness of Video-Feedback with Cognitive Preparation in Improving Social Performance and Anxiety through Super Skills for Life Programme Implemented in a School Setting. Int J Environ Res Public Health. 2020 Apr 18;17(8):2805. doi: 10.3390/ijerph17082805. PMID 32325756
- See also: Super Skills for Life original program's webpage — https://www.superskillsforlife.com/